CLINICAL TRIAL: NCT05214742
Title: Developing Derived Induced Pluripotent Stem Cells From Blood as a Model for the Study to Understand Imprinted Disorders
Brief Title: Developing Derived Induced Pluripotent Stem Cells as a Model to Understand Imprinted Disorders
Acronym: ID-STEM
Status: Enrolling by invitation | Type: Observational
Sponsor: Institute of Cardiometabolism and Nutrition, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A01597-34
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-01

CONDITIONS: Induced Pluripotent Stem Cells

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Silver-Russell Syndrome
  Interventions: Other: Diagnostic Test
- Beckwith-Wiedemann Syndrome
  Interventions: Other: Diagnostic Test
- Temple Syndrome
  Interventions: Other: Diagnostic Test

INTERVENTIONS:
Other: Diagnostic Test — Molecular diagnosis carried out in the context of care

SUMMARY:
Fetal and postnatal growth is finely regulated by genetic, epigenetic and environmental mechanisms. Parental imprinting is a regulatory mechanism that allows monoallelic expression of certain genes from a single parental allele through differential DNA methylation. Imprinted genes play a very important role in the control of fetal and postnatal growth. The pathophysiological mechanisms of these epimutations are largely unknown.

Studying the consequences of these epimutations on the molecular signature of the imprinted gene network in these patients would provide a better understanding of the epigenetic mechanisms regulating fetal growth. As these genes are weakly expressed in fibroblasts, these studies will be carried out on pluripotent stem cells or IPSCs (Induced Pluripotent Stem Cells).

ELIGIBILITY:
Inclusion Criteria:

1. Minor or young adult patients treated in the department, suffering from rare growth diseases: Silver-Russell syndrome (SRS), Beckwith-Wiedemann syndrome (BWS) and Temple syndrome (TS)
2. For minors, the patient's weight must be ≥ 5 kg

Exclusion Criteria:

* Patients unable to express their opposition to the use of their personal data.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: During their follow-up visit, parents and patients who meet the inclusion criteria will be asked to participate in the study. In the case of minors, their personal adhesion will be sought if their capacity of comprehension allows it after adapted written information.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-01-19 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The objective of the study is to understand the consequences of epimutations found | 1 day
  The objective of the study is to understand the consequences of epimutations found at 11p15 or 14q32 in these three syndromes (SRS, BWS and TS) on the network of genes subject to parental imprinting, in order to progress in the understanding of the mechanisms governing the epigenetic regulation of fetal growth.

CONTACTS AND LOCATIONS:
Overall Officials: Irène NETCHINE, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Hôpital Trousseau, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
IPD will be sahred with partners
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Access Criteria: Partners